CLINICAL TRIAL: NCT01868841
Title: 123-I mIBG (AdreView) Heart-to-Mediastinal (H/M) Ratio and SPECT Imaging
Brief Title: 123-I mIBG (AdreView) Heart-to-Mediastinal (H/M) Ratio and SPECT Imaging on a Small Field of View-High Efficiency Cardiac SPECT System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Timothy M. Bateman (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor-Investigator, Timothy M. Bateman, Medical Director, Aspire Foundation
Organization: Aspire Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-039
Record Dates: First submitted 2013-05-14; First posted 2013-06-05 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure; Cardiomyopathy
Keywords: 123I-mIBG; AdreView; SPECT; Heart to Mediastinal Ratio
MeSH Terms: conditions — Heart Failure; Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adreview LFOV SPECT Imaging followed by SFOV-HE Imaging (Active Comparator): SPECT imaging of 10 millicurie of Adreview
  Interventions: Drug: AdreView; Other: Single Photon Emission Computed Tomography
- AdreView SFOV-HE SPECT Imaging followed by LFOV Imaging (Active Comparator): SPECT imaging of 10 millicurie of Adreview
  Interventions: Drug: AdreView; Other: Single Photon Emission Computed Tomography

INTERVENTIONS:
Drug: AdreView — 10 millicurie of AdreView (123I-mIBG)
Other: Single Photon Emission Computed Tomography
  Other Names: SPECT

SUMMARY:
The purpose of this study is to demonstrate correlation of the H/M ratio of AdreView when derived from a large field of view Anger SPECT system and from a small field of view high sensitivity (CZT) SPECT system.

ELIGIBILITY:
Inclusion Criteria:

* New York Heart Association Class II or III Heart Failure
* Left ventricular ejection fraction less than or equal to 35%

Exclusion Criteria:

* Uncompensated heart failure
* Recent hospitalization within 30 days of cardiac related indications

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-12; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Relationship of H/M ratios obtained on LFOV and SFOV-HE systems | 3 months post-enrollment close
  H/M ratios as described will be calculated for the LFOV, and SFOV-HE data sets to determine the correlation between the two measurements. The r value, slope and intercept of this correlation will constitute the primary endpoint of this study. Specifically, we will establish the r value, slope and intercept for: LFOV-Planar vs LFOV-TOMO, LFOV-Planar vs SFOV-HE-TOMO, LFOV-TOMO vs SFOV-HE-TOMO.

SECONDARY OUTCOMES:
Image Quality | 3 month post-enrollment close
  We will investigate differences between the measurements in the SFOV-HE using the forward projections of the tomographic data and tomographic measurements of the H/M as other methods of establishing the correlation between tomographic and planar measurement of mIBG uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M Bateman, MD, Principal Investigator — Aspire Foundation
Locations (1):
- Cardiovascular Imaging Technologies, Kansas City, Missouri, United States